CLINICAL TRIAL: NCT03767855
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Multi-Part, Single and Multiple Ascending Dose Study of CK-3773274 in Healthy Adult Subjects
Brief Title: A Single and Multiple Ascending Dose Study of CK-3773274 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: CY 6011
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2020-01

CONDITIONS: Symptomatic Obstructive Hypertrophic Cardiomyopathy; Healthy Subjects
Keywords: CK-3773274; CK-274; obstructive hypertrophic cardiomyopathy; oHCM; aficamten
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- CK-3773274 for SAD Cohorts (Experimental): Subjects will be assigned to one of 8 planned dose cohorts and receive single doses of CK-3773274
  Interventions: Drug: CK-3773274 - Granules in Capsule
- Placebo for SAD Cohorts (Placebo Comparator): Subjects will be assigned to one of 8 planned dose cohorts and receive single doses of placebo
  Interventions: Drug: Placebo - Granules in Capsule
- CK-3773274 for MAD Cohorts (Experimental): Subjects will be assigned to one of 3 planned dose cohorts and receive multiple doses of CK-3773274
  Interventions: Drug: CK-3773274 - Granules in Capsule
- Placebo for MAD Cohorts (Placebo Comparator): Subjects will be assigned to one of 3 planned dose cohorts and receive multiple doses of placebo
  Interventions: Drug: Placebo - Granules in Capsule
- CK-3773274 for CYP2D6 Cohort (Experimental): Subjects with CYP2D6 poor metabolizer phenotype will be assigned to receive a single dose of CK-3773274
  Interventions: Drug: CK-3773274 - Granules in Capsule
- Placebo for CYP2D6 Cohort (Placebo Comparator): Subjects with CYP2D6 poor metabolizer phenotype will be assigned to receive a single dose of placebo
  Interventions: Drug: Placebo - Granules in Capsule
- Food Effect (Experimental): Subjects will be administered CK-3773274 with and without food in a randomized cross-over fashion
  Interventions: Drug: CK-3773274 - Granules in Capsule
- Relative Bioavailability (Experimental): Subjects will be administered CK-3773274 as granules in a capsule and as a tablet in a randomized cross-over fashion.
  Interventions: Drug: CK-3773274 - Granules in Capsule; Drug: CK-3773274 - Tablets

INTERVENTIONS:
Drug: CK-3773274 - Granules in Capsule — CK-3773274 formulated as granules in capsule
  Arms: CK-3773274 for CYP2D6 Cohort; CK-3773274 for MAD Cohorts; CK-3773274 for SAD Cohorts; Food Effect; Relative Bioavailability
Drug: Placebo - Granules in Capsule — Placebo formulated as granules in capsule
  Arms: Placebo for CYP2D6 Cohort; Placebo for MAD Cohorts; Placebo for SAD Cohorts
Drug: CK-3773274 - Tablets — CK-3773274 formulated as tablets
  Arms: Relative Bioavailability

SUMMARY:
The purposes of this study are to:

1. Learn about the safety of CK-3773274 after a single dose and multiple doses in healthy subjects.
2. Learn how healthy subjects tolerate CK-3773274 after a single dose and multiple doses.
3. Find out how much CK-3773274 is in the blood after a single dose and multiple doses.
4. Determine the effect of doses of CK-3773274 on the pumping function of the heart.
5. Evaluate the effect of cytochrome genetic variants on how the body metabolizes CK-3773274.
6. Evaluate the effect of a meal on how much CK-3773274 is in the blood in healthy adult subjects.
7. Evaluate whether the amount of CK-3773274 in the blood is the similar for both the tablet and granules in capsule forms of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females (of non-childbearing potential) between 18 and 55 years of age, inclusive
2. Body weight > 55.0 kg and body mass index within 18.0 to 32.0 kg/m2, inclusive
3. Normal cardiac structure and function, or if abnormalities are present, they are deemed not clinically significant
4. Normal to high left ventricular ejection fraction.
5. Normal electrocardiogram (ECG) or, if abnormalities are present, they are deemed not clinically significant
6. Clinical laboratory findings within normal range
7. Negative hepatitis panel (including hepatitis B surface antigen and hepatitis C antibody), and negative human immunodeficiency virus antibody screens
8. Willing and able to refrain from strenuous exercise (eg, activity which could be expected to cause muscle soreness)
9. For Arms 5 and 6 only: Subject is a CYP2D6 poor metabolizer

Exclusion Criteria:

1. History of any significant illness or disorder
2. History of stomach or intestinal surgery or resection (appendectomy, hernia repair, and/or cholecystectomy will be allowed)
3. A clinically significant illness within 4 weeks of Check-in
4. Inability to swallow capsules or tablets
5. History of or current substance abuse (drug or alcohol), known drug or alcohol dependence within the last 2 years prior to Screening, or positive test for drugs of abuse during the screening period
6. Use of any tobacco-containing or nicotine-containing products within 3 months prior to Check-in
7. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 30 days prior to Check-in
8. Any blood donation within 60 days of dosing, plasma donation within 30 days of dosing, or receipt of blood products within 2 months prior to Check-in

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events and Safety Signals observed during single and multiple ascending doses of CK-3773274 administered orally to healthy adult subjects. | SAD Cohorts: Day -1 - Day 10; CYP2D6 Cohort: Day -1 - Day - 24; MAD Cohorts: Day -1 - Day 27; Food Effect Cohort: Day -1 - Day 24; relative Bioavailability Cohort: Day -1 - Day 29
  Subject incidence of AEs, SAEs, and reduced LVEF

SECONDARY OUTCOMES:
Cmax of CK-3773274 after single and multiple ascending doses | SAD Cohorts: Day 1; CYP2D6 Cohort: Day 1; MAD Cohorts: Day 14 or Day 17; Food Effect Cohort: Day 15; Relative Bioavailability Cohort: Day 15
  Maximum concentration after dosing (Cmax) following single and multiple doses of CK-3773274 administered to healthy subjects
Change in absolute reduction in ejection fraction relative to baseline with doses of CK-3773274 | Time Frame for SAD Cohorts: Day -1 - Day 10; Time Frame for CYP2D6 Cohort: Day -1 - Day 24; Time Frame for MAD Cohorts: Day -1 - Day 27
  Changes from baseline in LVEF as measured by echocardiography with doses of CK-3773274
Assess the effect of CYP2D6 genetic variants on the PK of CK-3773274 | Day -1 - Day 24
  Maximum concentration after dosing (Cmax) following a single dose administered to CYP2D6 poor metabolizers
Assess the effect of a meal on how much CK-3773274 is in the blood in healthy subjects | Day -1 - Day 24
  Maximum concentration after dosing (Cmax) following single and multiple doses of CK-3773274 administered to healthy subjects in fed and fasted states
Relative bioavailability of CK-3773274 formulated as granules in capsule versus a tablet in healthy adult subjects | Time Frame for Bioavailability Cohort: Day -1 - Day 29
  PK parameters such as AUC calculated using plasma concentrations of CK-3773274

CONTACTS AND LOCATIONS:
Overall Officials: Study Director MD, Study Director — Cytokinetics
Locations (1):
- Clinical Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malik FI, Robertson LA, Armas DR, Robbie EP, Osmukhina A, Xu D, Li H, Solomon SD. A Phase 1 Dose-Escalation Study of the Cardiac Myosin Inhibitor Aficamten in Healthy Participants. JACC Basic Transl Sci. 2022 Aug 10;7(8):763-775. doi: 10.1016/j.jacbts.2022.04.008. eCollection 2022 Aug. PMID 36061336